CLINICAL TRIAL: NCT00019838
Title: Phase I and Pharmacokinetic Study of UCN-01 and Fludarabine in Relapsed or Refractory Low-Grade Lymphoid Malignancies
Brief Title: UCN-01 and Fludarabine in Treating Patients With Recurrent or Refractory Lymphoma or Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067252; NCI-99-C-0127; NCI-T99-0022; NCT00001822 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2005-02

CONDITIONS: Leukemia; Lymphoma
Keywords: Waldenström macroglobulinemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — 7-hydroxystaurosporine; fludarabine phosphate

INTERVENTIONS:
Drug: 7-hydroxystaurosporine
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die. Combining UCN-01 with chemotherapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of fludarabine when given with UCN-01 in treating patients with recurrent or refractory low-grade lymphoma or leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and toxic effects of fludarabine when administered with UCN-01 in patients with recurrent or refractory low-grade or indolent lymphoid malignancies.
* Determine, preliminarily, the activity of this treatment regimen in these patients.
* Assess the pharmacokinetics of this treatment regimen in these patients.

OUTLINE: This is a dose-escalation study of fludarabine.

Patients receive UCN-01 IV over 72 hours on days 1-3 alone during course 1 and over 36 hours on days 1-2 during courses 2-7. Patients also receive fludarabine IV over 30 minutes beginning on day 1 and continuing for up to 5 days during courses 2-7. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of fludarabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 2 months for 6 months, every 3 months for 1 year, and then every 6 months thereafter.

PROJECTED ACCRUAL: Approximately 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent or refractory low-grade or indolent lymphoid malignancies requiring systemic therapy, including the following:

  * Grade I or II follicular small cleaved cell lymphoma
  * Small lymphocytic lymphoma/leukemia subtypes (chronic lymphocytic leukemia)
  * Mantle cell lymphoma
  * Waldenstrom's macroglobulinemia
  * Lymphoplasmacytoid
  * Marginal zone (nodal, extranodal, or splenic subtypes)
  * Hairy cell leukemia
* Transformed indolent subtypes allowed provided 1 of the following criteria are met:

  * Previously treated with a doxorubicin-containing regimen
  * No rapidly progressing disease that threatens vital functions
* Measurable disease
* No active leptomeningeal or parenchymal CNS lymphoma NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 50,000/mm^3
* No active Coomb's-positive hemolytic anemia

Hepatic:

* Total bilirubin less than 2.0 mg/dL (unless elevation is due to Gilbert's disease and direct bilirubin is normal)

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No angina
* No congestive heart failure
* No myocardial infarction within the past 6 months

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No insulin-dependent diabetes mellitus

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* More than 3 weeks since prior systemic chemotherapy and recovered

Endocrine therapy:

* More than 3 weeks since prior systemic steroid therapy and recovered

Radiotherapy:

* Not specified

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-07

CONTACTS AND LOCATIONS:
Overall Officials: Wyndham H. Wilson, MD, PhD, Study Chair — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland

REFERENCES:
- [Result] Marti GE, Stetler-Stevenson M, Grant ND, White T, Figg WD, Tohnya T, Jaffe ES, Dunleavy K, Janik JE, Steinberg SM, Wilson WH. Phase I trial of 7-hydroxystaurosporine and fludararbine phosphate: in vivo evidence of 7-hydroxystaurosporine induced apoptosis in chronic lymphocytic leukemia. Leuk Lymphoma. 2011 Dec;52(12):2284-92. doi: 10.3109/10428194.2011.589547. Epub 2011 Jul 12. PMID 21745173
- [Result] Wilson WH, Gutierrez M, Stetler-Stevenson M, et al.: Phase I trial of 7-hydroxystaurosporine (UCN-01) and fludararbine phosphate (FAMP); in vivo evidence of UCN-01 induced apoptosis in CLL. [Abstract] Blood 96 (11 Pt 1): A-3268, 756a, 2000.